CLINICAL TRIAL: NCT05499039
Title: High Flow Nasal Cannula Versus Non-Invasive (NIV)in Both Hypoxemic and Hypercapnic Respiratory Failure.
Acronym: Highflow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Alham, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HFNC VS NIV
Record Dates: First submitted 2022-03-07; First posted 2022-08-12 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Acute Hypoxemic Respiratory Failure; Acute Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: patients with will be randomly enrolled to either non invasive group or HFNC group and improvement and patient satisfaction will be assessed
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participant , care provider , the investigator nor the outcome assessor will select patients in both groups , see results of other patients till the end of the study or informed by literature opinion in this intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A1 (NIVMV on hypoxemic) (Active Comparator): Use of NIV on acute hypoxemic respiratory failure patients
  Interventions: Device: Non-Invasive Mechanical Ventilation (NIV)
- Group A2 (HFNC on hypoxemic) (Experimental): Use of HFNC on acute hypoxemic respiratory failure patients
  Interventions: Device: High flow nasal cannula (HFNC)
- Group B1 (NIVMV on hypercapneic) (Active Comparator): Use of NIV on acute hypercapneic respiratory failure patients
  Interventions: Device: Non-Invasive Mechanical Ventilation (NIV)
- Group B2 (HFNC on hypercapneic) (Experimental): Use of HFNC on acute hypercapneic respiratory failure patients
  Interventions: Device: High flow nasal cannula (HFNC)

INTERVENTIONS:
Device: High flow nasal cannula (HFNC) — High flow nasal cannula consists of an apparatus that allows adjustable FiO2 from 21 to 100% and delivers a modified gas flow up to 60 l/ min .
  will be set with: -
  Temperature at 37°C or 34°C Flow rate 30: 50 L/min. FiO2 will be adjusted to achieve a SpO2 at least 95%
  Other Names: High velocity nasal insufflation (vapotherm)
  Arms: Group A2 (HFNC on hypoxemic); Group B2 (HFNC on hypercapneic)
Device: Non-Invasive Mechanical Ventilation (NIV) — Respiratory assistance is provided by a NIV either Puritan Bennet 840 , Engström Carestation or Hamilton-G5 , will be used for conventional non-invasive ventilation via an oronasal mask. Settings will be adjusted based on the clinical assessment of the respiratory therapist . Initial setting includes: -
  Positive End Expiratory Pressure (PEEP): 5 cmH2O. Pressure support (PS): 12-20 cmH2O. FiO2 will be adjusted to achieve a SpO2 at least 95% Intervention: Device: non-invasive ventilation
  Arms: Group A1 (NIVMV on hypoxemic); Group B1 (NIVMV on hypercapneic)

SUMMARY:
high flow nasal cannula (HFNC) oxygen therapy utilizes an air oxygen blend allowing from 21 % to 1 00% FiO2 delivery and generates up to 60 L/min flow rates The gas is heated and humidified through an active heated humidifier and delivered via a single limb heated inspiratory circuit (to avoid heat loss and condensation) to the patient through a large diameter nasal cannula Theoretically, HFNC offers significant advantages in oxygenation and ventilation over COT. Constant high flow oxygen delivery provides steady FiO2 and decreases oxygen dilution. It also washes out physiologic dead space and generates positive end expiration pressure (PEEP) that augments ventilation The heated humidification facilitates secretion clearance, decreases bronchospasm, and maintains mucosal integrity.

This study aims to evaluate the effectiveness of HFNC compared to NIMV in management of Acute hypoxemic and acute hypercapneic respiratory failure

DETAILED DESCRIPTION:
* Acute respiratory failure (ARF) is a common and serious complication among hospitalized patients. It is the most frequent reason for admission to the intensive care unit (ICU) . It carries an in-hospital mortality rate of 20.6% and cost 54.3 billion dollars nationwide in United States in 2009. Among those patients with ARF, 42.1 % of patients require mechanical ventilation (MV), which is associated with a significant increase in both length of stay and medical expense
* ARF can be categorized into acute hypoxemic respiratory failure(AHRF) and acute hypercapneic respiratory failure.
* Supplemental oxygen and treatment of the underlying cause is the mainstay of therapy for AHRF. Options for oxygen therapy include conventional oxygen therapy delivered via nasal cannulae (NC) or face masks (FM) initially, followed by non-invasive ventilation (NIV), and finally intubation or mechanical ventilation (MV) .
* Traditional NC and FM (collectively referred to as conventional oxygen therapy or COT) can achieve flow rates of up to 1 5 L/min. However, these flow rates may be significantly lower than patients' spontaneous inspiratory flow rates and the oxygen is diluted as it is mixed with room air Consequently, the fraction of inspired oxygen (FiO2) delivered Is variable and this is thought to explain why many patients require an escalation of oxygen therapy to NIV or MV.
* By contrast, humidified high flow nasal cannula (HFNC) oxygen therapy utilizes an air oxygen blend allowing from 21 % to 1 00% FiO2 delivery and generates up to 60 L/min flow rates The gas is heated and humidified through an active heated humidifier and delivered via a single limb heated inspiratory circuit (to avoid heat loss and condensation) to the patient through a large diameter nasal cannula Theoretically, HFNC offers significant advantages in oxygenation and ventilation over COT. Constant high flow oxygen delivery provides steady FiO2 and decreases oxygen dilution. It also washes out physiologic dead space and generates positive end expiration pressure (PEEP) that augments ventilation The heated humidification facilitates secretion clearance, decreases bronchospasm, and maintains mucosal integrity
* HFNC has been well studied in the neonatal and pediatric settings However, in adults, the use of HFNC has Primarily been studied in post-cardiac surgery post-extubation and bronchoscopy patients. However, the utility of HFNC use in adults with AHRF in emergency and general inpatient practice is less clear .Heated and humidified high-flow oxygen through nasal cannula (HFNC) has been developed over the past 2 decades, as an alternative to standard oxygen delivery systems
* . In adults, it has been used to treat hypoxemic respiratory failure, cardiogenic pulmonary edema, postoperatively and postextubation in do-not-intubate patients or during bronchoscopy
* To date, the literature supports the possibility to use HFNC as alternative to non-invasive ventilation (NIV) in some settings, while in others might be even superior . It is also an alternative to standard oxygen as first line therapy in management of patients with acute respiratory failure . NIV is strongly recommended in patients with acute-on-chronic respiratory failure associated with acute respiratory acidosis, the vast majority of whom meet the criteria for Chronic Obstructive Pulmonary Disease (COPD) exacerbation
* Recently, Studies revealed no difference of the 30-day mortality and intubation rate between NIV and HFNC, in severe acute exacerbation of COPD with moderate, hypercapnic, acute respiratory failure. In a retrospective study, that suggeste that HFNC oxygen therapy was beneficial, even in respiratory failure Type 2, resulting in significant improvement of both oxygenation and hypercapnia. another study also indicated that HFNO leads to a flow-dependent reduction in PaCO2 in patients with stable hypercapnic COPD, due to a washout of the respiratory tract and a functional reduction in dead space
* Although cumulative evidence supports that HFNC is effective in patients with hypercapnia, randomized studies to compare HFNC vs. NIV in patients with acute, hypercapnic respiratory failure are missing. so the investigator conducting this prospective, randomized, controlled trial, involving patients admitted to the Emergency Department (ED), to compare the efficacy of HFNC versus NIV in the management of acute hypercapnic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Acute hypoxemic respiratory failure. (Participants admitted with acute hypoxemic respiratory with the following criteria:

RR> 25 breath/minute Use of accessory muscles of respiration, paradoxical breathing, thoracoabdominal asynchrony.

Hypoxemia evidenced by PaO2 / FiO2 ratio <300)

* Acute hypercapnic respiratory failure ((Participants admitted with acute hypercapneic respiratory with the following criteria:

pO2 less than 60 mm Hg (hypoxemia). pCO2 greater than 50 mm Hg (hypercapnia) with pH less than 7.35. Signs and symptoms of acute respiratory distress)

Exclusion Criteria:

* Patients with preprocedural or post-procedural settings (ex: surgery, bronchoscope) post- extubation,
* Patients with cancer or transplant patients,
* Patients less than 18 years old
* Patients with Heart failure patients
* Patients with renal failure patients
* Patients with hemodynamic instability
* Patients with central causes of hypercapnic respiratory failure
* Patients with disturbed conscious level
* Patients who refuse to participate in the study
* Indication for emergency endotracheal intubation
* Tracheotomy or other upper airway disorders
* Active upper gastrointestinal bleeding

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of HFNC and NIV in correction of Acidosis . | Baseline
  Evaluation of the effectiveness of HFNC VS NIV in correction of Acidosis through measurement of PH via arterial blood gases test (ABG).
  Evaluation of the effectiveness of HFNC in correction of Acidosis through measurement of PH via arterial blood gases test (ABG).
Evaluation of HFNC and NIV in correction of Hypercapnia. | Baseline
  Evaluation of the effectiveness of HFNC VS NIV in correction of Hypercapnia through measurement of PCO2 by mmHg via arterial blood gases test (ABG)
Evaluation of HFNC and NIV in management of Acute hypoxemic respiratory failure. | Baseline
  Evaluation of the effectiveness of HFNC VS NIV in management of Acute hypoxemic respiratory failure through measurement of PO2 via arterial blood gases test (ABG)
Evaluation of HFNC and NIV in correction of Hypoxemia. | Baseline
  Evaluation of the effectiveness of HFNC VS NIV in correction of Hypoxemia through measurement of O2 saturation by percentage % via pulse oximeter.
Endotracheal intubation rate. | Baseline
  needs escalation to invasive mechanical ventilation

SECONDARY OUTCOMES:
In hospital mortality. | one month
  death
duration of intervention | one month
  time needed for ventilatory support
hospital coast | one month
  effects on hospital coast
duration of ICU stay . | one month
  icu occupancy
development of complications | one month
  due to devices

CONTACTS AND LOCATIONS:
Overall Officials: Zein Al-abdeen Ah Sayed, professor, Study Director — Assiut University; Taghred SA Meshref, professor, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No